CLINICAL TRIAL: NCT06525857
Title: Observing Physiological Changes in Patients With Long-term Oxygen Therapy Via Optical and Accelerometry Signals
Brief Title: Observing Physiological Changes in Patients With Long-term Oxygen Therapy
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: STD0006706
Record Dates: First submitted 2024-06-25; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: LTOT — Patients with newly prescribed LTOT will be monitored for physiological changes

SUMMARY:
In this project, the investigators aim to assess changes of physiological parameters obtained non-invasively through PPG and accelerometry signals between before and during LTOT (long-term oxygen therapy) and investigate if those changes are different in patients with worsening frailty and/or improving quality of life.

For this, they will record optical (PPG) and accelerometry data via a datalogger on 40 patients undergoing LTOT and assess the PPG-derived physiological signals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-year-old, and
* Chronic respiratory disease including a) chronic obstructive pulmonary disease, b) interstitial lung disease, c) pulmonary hypertension, d) bronchiectasis, and
* Prescribed new LTOT due to a chronic respiratory disease with resting and/or exertional hypoxemia, and
* Able to speak/read/understand German or French, and
* Willing and able to understand and provide signed informed consent

Exclusion Criteria:

* Pregnant or lactating women, or
* Inability to follow the procedures/instructions of the study (e.g. due to language, psychological disorders, dementia, etc.), or
* Patients having a subordination link to the investigators, or
* Patients with isolated nocturnal oxygen therapy or LTOT prescription for a heart disease, sleep associated breathing disorder, neuromuscular disease or lung cancer, or
* Known participation in another human research project (ClinO/HRO) that may affect the objectives of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a respiratory disease and newly prescribed LTOT
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate changes from before and during LTOT | From 1 week before start of LTOT to 1 month after start of LTOT
  Record heart rate (BPM) to compare before and during LTOT
Respiratory rate changes from before and during LTOT | From 1 week before start of LTOT to 1 month after start of LTOT
  Record respiratory rate (breaths per minute) to compare before and during LTOT
SpO2 changes from before and during LTOT | From 1 week before start of LTOT to 1 month after start of LTOT
  Record SpO2 (%) to compare before and during LTOT

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Guler, PD Dr. med., Principal Investigator — Universitätsklinik für Pneumologie, Allergologie und klinische Immunologie, Inselspital Bern
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No